CLINICAL TRIAL: NCT00171990
Title: Efficacy and Safety of Oral Famciclovir in Patients With Active Recurrent Genital Herpes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFAM810AAU01
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Recurrent Genital Herpes
Keywords: genital herpes; herpes; famciclovir
MeSH Terms: conditions — Herpes Genitalis; Herpes Simplex | interventions — Famciclovir

INTERVENTIONS:
Drug: Famciclovir

SUMMARY:
This is a phase III, multicenter, randomized, double-blind, parallel-group study to compare the efficacy and safety of a two-day treatment with famciclovir (500 mg loading dose followed by 250 mg 12-hourly) to standard five-day treatment with famciclovir (125 mg 12-hourly) in patients with active recurrent genital herpes.

This study is not recruiting patients in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of genital herpes
* Had at least 2 recurrences in past 12 months or 1 recurrence in past 6 months

Exclusion Criteria:

* - Currently taking suppressive herpes antiviral therapy
* Females who are pregnant, breast feeding or planning to become pregnant during study
* History of allergy to famciclovir or similar products (e.g. aciclovir, valaciclovir)

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1461 (Actual)
Dates: Start 2003-01; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Estimated probability being not lesion-free(i.e. not healed) 5.5 elapsed days (132 hours) after patient self-initiation therapy.

SECONDARY OUTCOMES:
Safety and tolerability assessed by AEs.
Time between recurrences of genital herpes.
Proportion of aborted (i.e. lesions did not appear)genital herpes recurrences. Change from baseline in symptoms or impairment. Change form baseline in functioning or disability.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, North Ryde, Australia